CLINICAL TRIAL: NCT00978978
Title: Propofol Versus Midazolam and Fentanyl for Diagnostic and Screening Colonoscopy in Patients With Advanced Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Jorge-Shmuel Delgado, MD., Department of Gastroenterology & Hepatology. Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SOR484909CTIL
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-09

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Fentanyl; Endoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol, endoscopies, liver diseases (Active Comparator): Propofol, endoscopies, liver diseases
  Interventions: Drug: Propofol VS. midazolam and fentanyl, endoscopies, liver diseases
- midazolam and fentanyl, endoscopies, liver diseases (Active Comparator): Control: midazolam and fentanyl, endoscopies, liver diseases
  Interventions: Drug: Propofol VS. midazolam and fentanyl, endoscopies, liver diseases

INTERVENTIONS:
Drug: Propofol VS. midazolam and fentanyl, endoscopies, liver diseases — 1. Intervention group (Propofol): It will be administered as a monotherapy under direct gastroenterologists'
  2. Control group (Midazolam with or without Fentanyl): Both drugs will be administered by the gastroenterologists

SUMMARY:
Prospective, randomized-controlled trial (RCT) comparing the use of Propofol and traditional sedation (Midazolam and Fentanyl) for diagnostic and screening endoscopies in patients with liver diseases. The investigators' working hypothesis is that the use of propofol will be translated in a shorter recovery and discharge times with a higher patient satisfaction and a decrease in general complications in the context of patients with advanced liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients older than 18 and younger than 75 years with advanced liver disease, defined by the presence of liver fibrosis at least F3 and higher in the METAVIR score or with established cirrhosis (Child Pugh A, B and C)

Exclusion Criteria:

* Patients with significant cardiorespiratory disease i.e. advanced respiratory, renal and heart failure (ASA class III or higher except for patients with decompensate liver cirrhosis), obstructive sleep apnea or those with mild degree of liver fibrosis (less than F3)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of propofol in liver diseases | At the end of each endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology. Soroka University Medical Center, Beersheba, Beer-Sheva, Israel